CLINICAL TRIAL: NCT05915091
Title: Comparative Effects of Dry Needling and Cross Friction Massage on Patients With Plantar Fascitis, a Randomized Controlled Trial
Brief Title: Comparative Effects of Dry Needling and Cross Friction Massage on Patients With Plantar Fascitis, RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/544
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental)
  Interventions: Diagnostic Test: Dry Needling
- Cross Friction Massage (Other)
  Interventions: Other: Cross Friction Massage

INTERVENTIONS:
Diagnostic Test: Dry Needling — Dry needling is a treatment that healthcare providers use for pain and movement issues associated with myofascial trigger points. With this technique, a provider inserts thin needles into or near your trigger points. The needles stimulate your muscles, which causes them to contract or twitch
  Arms: Dry Needling
Other: Cross Friction Massage — Cross friction massage breaks down scar tissue and remodels the tissue into more flexible, pliable, and functional, healthy soft tissue. Also known as transverse friction massage, this technique is a deep tissue massage technique performed at the site of injury
  Arms: Cross Friction Massage

SUMMARY:
Effectiveness Comparative Effects of Dry Needling and Cross Friction Massage on Patients With Plantar Fascitis

ELIGIBILITY:
Inclusion Criteria:

* Patients With Plantar Fascitis

Exclusion Criteria:

* Other Health Issues

Ages: 35 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain Scale of Plantar Fasciitis | 3 Months
Foot Health Status Questioner Score | 3 Months
Foot Function Index Score | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan